CLINICAL TRIAL: NCT00740844
Title: Evaluation of Intermittent Pneumatic Compression (IPC) of the Lower Limbs Associated With Elastic Stockings (ES) Compared to ES Alone on Venous Thromboembolism Incidence in Patients With High Bleeding Risk Hospitalized in Intensive Medical Care Units
Brief Title: Efficacy of Intermittent Pneumatic Compression (IPC) on Venous Thromboembolism Incidence in Intensive Care Unit (ICU) Patients With High Bleeding Risk
Acronym: CIREA1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Brest (Other)
Collaborators: Tyco Healthcare Group (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CIREA 1
Record Dates: First submitted 2008-08-22; First posted 2008-08-25 (Estimated); Last update posted 2025-12-03 (Actual); Status verified 2012-02

CONDITIONS: High Bleeding Risk; Hemorrhage
Keywords: Intermittent pneumatic compression; Hospitalization; Intensive care unit; High bleeding risk; Venous thromboembolism prophylaxis
MeSH Terms: conditions — Hemorrhage

ARMS (2):
- 1 (No Intervention): No intermittent pneumatic compression of the lower limbs during patient hospitalisation in réanimation unit
- 2 (Experimental): Intermittent pneumatic compression of the lower limbs during hospitalisation in reanimation unit
  Interventions: Device: Intermittent pneumatic compression of the lower limbs

INTERVENTIONS:
Device: Intermittent pneumatic compression of the lower limbs — Intermittent pneumatic compression of the lower limbs during hospitalisation in reanimation unit
  Arms: 2

SUMMARY:
This multicentre open-label randomized parallel-group trial aims to evaluate the association intermittent pneumatic compression + elastick stockings versus elasting stockings alone on symptomatic or asymptomatic venous thromboembolism incidence, evaluated systematically at day 6 (+/-2days), in patients hospitalized in intensive care units and with high bleeding risk.

DETAILED DESCRIPTION:
Background: Venous thromboembolism is a leading cause of morbi-mortality for patients hospitalized in intensive medical care units. Nevertheless, few studies evaluating prophylactic methods exist. Data from these studies demonstrate however that unfractionated heparin and low molecular weight heparin are effective to reduce the incident rate of asymptomatic deep venous thrombosis (DVT) of the lower limbs by 50 % compared to the absence of prophylaxis. Rate of asymptomatic DVT remains about 15 %. When the bleeding risk is high, drug prophylaxis with anticoagulants is contra-indicated, and mechanical devices are recommended: elastic stockings (ES) alone or associated with intermittent pneumatic compression (IPC). However, mechanical devices have not been systematically evaluated in intensive medical care units.

Objective:

To compare the association IPC + ES to ES alone in patients with high bleeding risk and hospitalized in intensive medical care units, on symptomatic or asymptomatic venous thromboembolism incidence, evaluated systematically at day 6.

Design: Multicentre open-label randomized parallel-group trial with blinded evaluation of outcomes, and an inclusion period of 24 month. Brest CIC (Centre d'Investigations Cliniques, research center) coordinates this multicentre trial.

Outcomes:

The primary endpoint is a combined criterion (blindly evaluated) between day 1 and day 6:

1. Non fatal symptomatic venous thromboembolic event (objectively confirmed) between day 1 and day 6,
2. death due to a pulmonary embolism between day 1 and day 6, and 3) asymptomatic DVT (distal or proximal) detected by ultrasonography systematically done at day 6.

Patients number:

CIREA 1 : Assuming a DVT frequency of 15 % in the control group (ES alone) , we calculated that 356 patients will be required for the study to have 80% power to detect a 60% reduction in the relative risk with a two-sided alpha level of 5%. Because of about 20 % deaths in the first days, we decide to increase the number at 392 subjects.

Statistical analysis: Efficacy analysis is performed on an 'intention-to-treat' basis. The frequencies of the combined primary outcome at day 6 are compared between groups using an exact one-sided Fischer test. Adjustment for stratification variables used Cochran-Mantel-Haenszel test. Relative risk and absolute risk reduction are computed with their 95% CIs. A logistic regression model is used to take into account potential imbalance in baseline characteristics.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 Years,
* Admission in intensive medical care unit
* High risk for hemorrhage
* Written informed consent given by the patient or relative.

High risk for hemorrhage is defined by:

* symptomatic bleeding or organic lesions likely to bleed,
* hemophilic diseases,
* haemostatic abnormalities: platelet count < 50 000/mm 3, APTT > 2 N, prothrombin time < 40%,
* recent intra-cerebral hemorrhage,
* severe anemia (Hemoglobin < 7 g/dl) due to a bleeding or unexplained.

Exclusion Criteria:

* Age < 18 years,
* Patient refusal,
* No high risk for hemorrhage
* Admission in intensive care unit ≥ 36 hours
* Admission in intensive care unit likely for < 72 hours
* A "do not resuscitate" order
* IPC contra-indication: Recent DVT (< 3 month), severe lower limbs arteriopathy (III and IV), any arterial graft of the legs, a wound in the lower limb related either to a vascular disease (ulcer) or a trauma.
* Patient with mechanical prosthetic heart valve.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 408 (Actual)
Dates: Start 2007-11; Primary Completion 2011-01 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Combined criterion evaluated at day 6 ± 2 days after randomization:symptomatic venous thromboembolic event, non fatal, objectively confirmed,Death related to PE,Asymptomatic DVT of the lower limbs detected by CUS on day 6 ± 2 days. | 6 days (+/- 2 days)

SECONDARY OUTCOMES:
Symptomatic thromboembolic events occurred between day 6 and day 90, and total mortality at 1 month and 3 months. | 6 days to 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Karine LACUT, MD, Study Director — CHU Brest France, Univ Brest, EA 3878
Locations (10):
- France (10):
  - Medical intensive care unit, Angoulême
  - HIA Clermont-Tonnerre, Brest
  - Medical Intensive Care Unit, Brest
  - Medical Intensive Care Unit, Lille
  - Intensive Care Unit, Limoges
  - Medical Intensive Care Unit, Nantes
  - Medical intensive care unit, Orléans
  - Medical Intensive Care Unit, Paris
  - Medical intensive care unit, Poitiers
  - Medical intensive care unit, Tours

REFERENCES:
- [Result] Vignon P, Dequin PF, Renault A, Mathonnet A, Paleiron N, Imbert A, Chatellier D, Gissot V, Lheritier G, Aboyans V, Prat G, Garot D, Boulain T, Diehl JL, Bressollette L, Delluc A, Lacut K; Clinical Research in Intensive Care and Sepsis Group (CRICS Group). Intermittent pneumatic compression to prevent venous thromboembolism in patients with high risk of bleeding hospitalized in intensive care units: the CIREA1 randomized trial. Intensive Care Med. 2013 May;39(5):872-80. doi: 10.1007/s00134-013-2814-2. Epub 2013 Jan 31. PMID 23370827